CLINICAL TRIAL: NCT04108013
Title: A Randomized,Controlled,Open-label,Prospective,Single-center Study to Investigate the Neoadjuvant Therapy of SHR-1210 in Combination With Carboplatin and Paclitaxel-albumin in Combination With Carboplatin and Paclitaxel in Resectable NSCLC
Brief Title: A Study of SHR-1210 in Combination With Carboplatin+Paclitaxel-albumin in Subjects With Resectable NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, zhangyi, Chief physician, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XWh-NSCLC-NEO-IIT-SHR1210
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Lung Cancer Stage II; PD-1 Antibody; Non-small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210+Carboplatin+Paclitaxel-albumin (Experimental): Subject will receive SHR-1210 200mg every 3 weeks, carboplatin AUC 5 on Day 1 of each 21 day, Paclitaxel-albumin 130mg/m2 on Day 1 and Day 8 of each 21 day, 2 cycles.
  Interventions: Drug: SHR-1210
- Carboplatin+Paclitaxel-albumin (Active Comparator): Subject will receive carboplatin AUC 5 on Day 1 of each 21 day, Paclitaxel-albumin 130mg/m2 on Day 1 and Day 8 of each 21 day, 2 cycles.
  Interventions: Drug: Carboplatin and Paclitaxel-albumin

INTERVENTIONS:
Drug: SHR-1210 — In the experimental group, 200mg SHR-1210 was given in the first day of each cycle, Carboplatin was given in the first day of each cycle, Paclitaxel-albumin was given in the first and eighth day of each cycle, with intravenous drip.
  Arms: SHR-1210+Carboplatin+Paclitaxel-albumin
Drug: Carboplatin and Paclitaxel-albumin — In the control group, Carboplatin was given in the first day of each cycle, Paclitaxel-albumin was given in the first and eighth day of each cycle, with intravenous drip.
  Arms: Carboplatin+Paclitaxel-albumin

SUMMARY:
This study is a randomized, controlled, open-label, prospective, single-center phase II clinical study. Target population is patients with stage II and IIIA resectable non-small cell lung cancer who had not received systemic chemotherapy. Study objective is to evaluate the major pathologic response of SHR-1210 + carboplatin + paclitaxel-albumin in subjects with resectable non-small cell lung cancer. SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
In this study, eligible subject will be randomized into study arm or control arm to accept study treatment. Subjects who randomized into control will have the opportunity to receive the treatment of carboplatin + paclitaxel-albumin therapy after confirmed disease progression. Treatment cycles of chemotherapy will be 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-70 years of age.
2. ECOG performance status of 0 or 1.
3. Life expectancy ≥ 12 weeks.
4. Subjects are diagnosed with histologically or cytologically confirmed NSCLC.
5. Subjects are diagnosed with resectable stage II, stage IIIA non-small cell lung cancer.
6. Subjects enrolled must have measurable lesion(s) according to the RECIST 1.1 standard (the CT scan length of the tumor lesion > 10 mm, the short diameter of CT scan of the lymph node lesions > 15 mm).
7. Subjects haven't received radiotherapy, chemotherapy, surgery and targeted therapy before admission.
8. Subjects must have adequate pulmonary function for expected pneumonectomy.
9. The main organ's function is normal and it should meet the following criteria:

(1)Blood routine examination should be complied with (No blood transfusion, no use of hematopoietic factors and no use of drugs for correction within 14 days):

a.ANC ≥ 1.5×109/L； b.HB ≥ 90 g/L； c.PLT ≥ 100×109/L；

(2)Biochemical tests must meet the following criteria:

1. TBIL ≤ 1.5ULN；
2. ALT、AST≤ 2.5 ULN (If abnormal liver function is caused by liver metastasis, ALT、AST< 5ULN;
3. sCr≤1.5ULN，endogenous creatinine clearance rate≥50ml/min(Cockcroft-Gault formula);

   (3)Blood coagulation must meet the following criteria: INR≤1.5 and APTT≤1.5 ULN；

   10.Women of childbearing age must undergo a serological pregnancy test within 3 days before the first dose with negative results and willing to use a medically approved and effective contraceptive method (e.g. intrauterine device, contraceptive pill or condom) during the study and within three months after the last dose. For male subjects whose partners are women of childbearing age, they should be sterilized surgically or agree to use effective contraceptive methods during the study and within three months after the last dose.

   11.Subjects should be voluntarily participate in clinical studies and informed consent should be signed.

   Exclusion Criteria:
   1. Subjects have symptomatic central nervous system metastasis.
   2. Subjects have a history of any active autoimmune disease or autoimmune disease including but not limited to the following: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism which can be included after hormone replacement therapy; Subjects with childhood asthma have been completely alleviated and without any intervention or vitiligo in adulthood can be included. Subjects who need medical intervention with bronchodilators can not be included.
   3. Subjects with congenital or acquired immunodeficiency such as HIV infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody is positive and HCV-RNA is higher than the lower detection limit of the analysis method) or co-infection with hepatitis B and hepatitis C.
   4. Subjects used immunosuppressive drugs excluding nasal spray and inhaled corticosteroids or systemic steroids at physiological doses(prednisolone≤10 mg/day or other corticosteroids of the same pharmacophysiological dose) within 14 days before the first dose.
   5. Subjects were vaccinated with live attenuated vaccine within 4 weeks before the first dose or during the study period.
   6. Subjects has taken last systemic cytotoxic or radiotherapy treatment in the past 4 weeks or subjects are currently using other antineoplastic drugs.
   7. Subjects suffered from other malignant tumors in the past three years.
   8. There is evidence that subjects have pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-induced pneumonia and severe impairment of lung function.
   9. Subjects have uncontrollable hypertension (systolic pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg), despite patients have taken the best drug treatment;
   10. Subjects with grade II or above myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (QTc interval > 450 ms for males and QTc interval < 470 ms for females). Subjects with grade III-IV cardiac insufficiency or with left ventricular ejection fraction (LVEF) less than 50% had myocardial infarction within 6 months before admission according to NYHA criteria. Subjects with grade II or above heart failure, uncontrolled angina, uncontrolled severe ventricular arrhythmias, clinically pericardial disease, acute ischemia or abnormal active conduction system.
   11. The subjects developed severe infection within 4 weeks before the first dose (such as: intravenous antibiotics, antifungal or antiviral drugs), or fever of unknown reason (>38.5 °C) before the first dose or during the first screening period.
   12. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation is known.
   13. Pregnant or lactating women; Fertile subjects who are unwilling or unable to take effective contraceptive measures
   14. It is known that subjects have allergic reaction, hypersensitivity reaction or intolerance to SHR-1210, paclitaxel-albumin or its excipients.
   15. Investigators believe that there is any situation that could damage the subjects or cause the subjects to fail to meet or perform the research requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-10-08 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 3.5 months
  It is defined as residual tumors less than 10% after neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Objective Response Rate | 6.5 months
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.
Pathological complete response | 3.5 months
  No histologic evidence of malignancy or only the ingredients of carcinoma in situ was found in primary tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Doctor, Principal Investigator — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No